CLINICAL TRIAL: NCT01624116
Title: A Comparison of Four Hypoglycaemic Regimens During Ramadan Fasting in Type 2 Diabetic Patients and the Effect of Add-On Acarbose on Glycaemic Excursions During Ramadan Fasting
Brief Title: Comparison of Hypoglycaemic Regimens During Ramadan Fasting in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Services Hospital, Lahore (Other Government)
Responsible Party: Principal Investigator, Dr Saira Burney, Senior Registrar, Endocrinology Unit & Diabetes Management Centre, Services Institute of Medical Sciences,Lahore,Pakistan., Services Hospital, Lahore
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RT2011
Record Dates: First submitted 2012-03-19; First posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Diabetes, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Acarbose; Diet; Metformin; glimepiride; Sitagliptin Phosphate, Metformin Hydrochloride Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Diet and lifestyle measures alone. (Active Comparator): Type 2 diabetic subjects on lifestyle counselling as part of diabetes treatment would continue as such during Ramadan. They would receive acarbose on one day to be followed by CGMS for a 24 hour period
  Interventions: Drug: Acarbose; Other: Diet and lifestyle
- Metformin monotherapy (Active Comparator): Type 2 diabetics on biguanide treatment.
  Interventions: Drug: Acarbose; Other: Diet and lifestyle; Drug: Metformin
- Metformin + Sulphonylurea. (Active Comparator): Type 2 diabetics on dual oral hypoglycaemics-metformin and glimepiride.
  Interventions: Drug: Acarbose; Other: Diet and lifestyle; Drug: Metformin/ Glimepride
- Metformin + Sitagliptin (Active Comparator): Type 2 diabetics managed on dual oral hypoglycaemic therapies: metformin and sitagliptin.
  Interventions: Drug: Acarbose; Other: Diet and lifestyle; Drug: Metformin/Sitagliptin

INTERVENTIONS:
Drug: Acarbose — Tab.Acarbose 50mg BD for one day in addition to existing medication to 10% of patients in each treatment arm.
  Other Names: *Tab.Glucobay 50mg (Bayer).
Other: Diet and lifestyle — Patients would follow a 1200 KCal Ramadan diet plan, and exercise for 30 minutes per day
Drug: Metformin — Patients on metformin monotherapy prior to Ramadan will continue on it, in the same dose
  Other Names: Tablets Glucophage (Merck)
  Arms: Metformin monotherapy
Drug: Metformin/ Glimepride — Metformin 500mg and Glimepride 1mg in a combination tablet. Dosage frequency BD
  Other Names: Tablet Getformin 1/500 (Getz Pharma)
  Arms: Metformin + Sulphonylurea.
Drug: Metformin/Sitagliptin — Metformin 500 and sitagliptin 50mg in a combination tablet,dosage frequency BD.
  Other Names: Tab.TreviaMet 50/500 (Getz Pharma)
  Arms: Metformin + Sitagliptin

SUMMARY:
Type 2 diabetic patients who fast during Ramadan experience swings in glycaemic control between hypoglycaemic troughs and hyperglycaemic spikes. Hence, the dual challenge in fasting diabetics is to identify which treatment modality leads to the most stable blood glucose levels during a fast and how to smooth out these excursions and reduce risks of fast to a minimum.

DETAILED DESCRIPTION:
Study Objectives:

* To compare changes in clinical and metabolic parameters from baseline to the end of four weeks fasting in Ramadan between four treatment arms:

  * diet and lifestyle measures alone.
  * metformin monotherapy.
  * combination therapy with metformin + sulfonylurea.
  * combination therapy with metformin + sitagliptin.
* To compare the 24 hour CGMS profile during Ramadan fasting in type 2 diabetic patients before and after addition of acarbose to these pre-existing sub-maximal hypoglycaemic regimens.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c 6.5-9.5%.
* Type 2 diabetics on two or less oral hypoglycaemic agents.

Exclusion Criteria:

* Any contraindications either to fasting or to any of the trial medication.
* Pregnancy.
* Serum creatinine > 1.4 mg/dl.
* Serum ALT > twice upper limit normal.
* History of pancreatitis, serum amylase > twice upper limit normal.
* History of intolerance to acarbose.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2011-08; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Change in body weight and fructosamine levels during Ramadan fasting. | 28 days (Average duration of Ramadan fasting)
  Change in body weight and fructosamine levels from baseline to end of Ramadan.

SECONDARY OUTCOMES:
Change in fasting lipid profile from baseline to end of Ramadan. | 28 days(average duration of Ramadan)
  Change in fasting lipid profile from baseline to end of Ramadan.
Change in ghrelin levels from baseline to end of Ramadan. | 28days (average duration of Ramadan)
  Change in ghrelin levels from baseline to end of Ramadan.
Change in renal profile from baseline to end of Ramadan | 28 days(average duration of Ramadan)
  Change in renal profile from baseline to end of Ramadan.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Khadija Irfan, MBBS,FCPS, Principal Investigator — Services Hospital.
Locations (1):
- Endocrinology Unit & Diabetes Management Centre, Services Hospital., Lahore, Pakistan